CLINICAL TRIAL: NCT07119632
Title: Clinical Study Plan of Medicine Stick Therapy Combined With Repeated Urotong Therapy on Lower Limb Dysfunction in Patients With Stroke
Brief Title: Study of Medicine Stick Therapy Combined With Repeated Urotong Herapy on Lower Limb Dysfunction in Stroke Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jiangen Ye (Other)
Responsible Party: Sponsor-Investigator, Jiangen Ye, associate professor, Second Affiliated Hospital of Nanchang University
Organization: Second Affiliated Hospital of Nanchang University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2024B0564
Record Dates: First submitted 2025-07-09; First posted 2025-08-13 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Medication stick therapy +Repetitive facilitative exercise (Experimental): 1. Medication stick therapy:The specific operation is as follows: The patient lies down, holds the rods with both hands, and massages and squeezes the muscles from the muscle end towards the starting end while applying the medicinal wine. This causes the muscles to contract in a centripetal direction. The treatment is considered successful when there is local heat and the skin becomes flushed. It is performed 20 minutes per time, once a day, 6 times a week, for a total of 6 weeks.
  2. Repetitive facilitative exercise: It includes specific movement patterns of the affected lower limb and weight-bearing training on the healthy side.Each movement pattern is performed 100 repetitions with the therapist's assistance, once a day, 6 days a week, for a total of 6 weeks of continuous treatment.
  Interventions: Other: RFE therapy
- Repetitive facilitative exercise (Active Comparator): Repetitive facilitative exercise: It includes specific movement patterns of the affected lower limb and weight-bearing training on the healthy side.Each movement pattern is performed 100 repetitions with the therapist's assistance, once a day, 6 days a week, for a total of 6 weeks of continuous treatment.
  Interventions: Other: RFE therapy

INTERVENTIONS:
Other: RFE therapy

SUMMARY:
At present, domestic scholars have applied medicine stick therapy and repetitive facial exercise (RFE) to the rehabilitation treatment of stroke patients, but there are few relevant literature reports on medicine stick therapy combined with RFE and show the differences in the effects of the two different treatment methods. To this end, this study intends to follow up the effects and effects of drug stick therapy and its combined effect with RFE on the recovery of lower limb motor function in patients after stroke, and follow up the patients' limb motor function, daily life activity ability, quality of life, balance function, etc.

DETAILED DESCRIPTION:
At present, domestic scholars have applied medicine stick therapy and repetitive facial exercise (RFE) to the rehabilitation treatment of stroke patients, but there are few relevant literature reports on medicine stick therapy combined with RFE and show the differences in the effects of the two different treatment methods. To this end, this study intends to follow up the effects and effects of drug stick therapy and its combined effect with RFE on the recovery of lower limb motor function in patients after stroke, and follow up the patients' limb motor function, daily life activity ability, quality of life, balance function, etc.; use the Fugl-Meyer motor function evaluation scale, Barthel index, Brunnstrom grading, Holden walking function and other scales to conduct multi-angle evaluation of stroke patients, combine traditional Chinese medicine rehabilitation with Western medicine rehabilitation treatment, combine these two different treatment technologies, give full play to their respective advantages and integrated effects to verify. The specific research content includes: participant recruitment and screening, random grouping design, baseline evaluation, treatment intervention, post-treatment evaluation, data statistics and analysis. This study aims to explore the feasibility and advantages of the combined application of drug stick therapy combined with RFE to provide more effective treatment methods for rehabilitation of stroke patients.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of stroke
* The first onset and the disease duration must be less than 3 months. exclusion criteria：
* Combined with other serious diseases such as severe cardiovascular, respiratory failure, liver and renal function damage, malignant tumors, etc.
* Consciousness disorders and cognitive impairment;
* Eczema, inflammation, infection, and scars at acupuncture points or skin;

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Modified Barthel Index | From enrollment to 8 weeks of treatment
  The Modified Barthel Index has a minimum score of 0 and a maximum score of 100. The higher the score, the better the functional ability.

SECONDARY OUTCOMES:
Holden Walking Function | From enrollment to 8 weeks of treatment
  Holden Walking Function: Minimum level 0, maximum level 6. The higher the level, the better the function.

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2025-01-18): https://cdn.clinicaltrials.gov/large-docs/32/NCT07119632/ICF_000.pdf